CLINICAL TRIAL: NCT01950715
Title: Evaluation of the Gastro-colic Response in IBS Patients Treated With Sacral Nerve Stimulation
Brief Title: Multimodal Stimulation Before and After Sacral Nerve Stimulation for Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201302, JLF
Record Dates: First submitted 2013-09-12; First posted 2013-09-25 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Sacral Nerve Stimulation; Gastro-colic response; Multimodal Stimulation
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sacral nerve stimulation (Other): A single armed study to evaluate the on the gastro-colic response in IBS patients treated with sacral nerve stimulation
  Interventions: Device: sacral nerve stimulation

INTERVENTIONS:
Device: sacral nerve stimulation — Sacral nerve stimulation
  Other Names: External pacemaker, model 3625, Medtronic Inc.

SUMMARY:
Sacral nerve stimulation (SNS) has become a well-established treatment for patients with fecal incontinence since 1995. The mechanism of action of SNS is still not fully understood but recent studies have shown changes in both colonic motility and rectal sensibility. The investigators have previously shown IBS patients to benefit from sacral nerves stimulation. With the present study, the investigators aim to evaluate if sacral nerve stimulation alters the gastro-colic response in IBS patients.

DETAILED DESCRIPTION:
Twenty four patients with IBS-D or IBS-M according to the ROME III criteria, will be enrolled in the study.

Having meet inclusion criteria, the patients will be examined with Multimodal Stimulation at baseline and at six weeks in the sacral nerve stimulation test period.

During the Multimodal Stimulation the patients will have impedance planimetry conducted before and after a standardised meal to evaluate on their gastro-colic response without and during sacral nerve stimulation.

The patients enrolled in the study will in the same time period participate in another study evaluating subsensory sacral nerve stimulation. A study registered at clinical trials.

Here patients are randomised to receive either OFF-subsensory or subsensory-OFF stimulation in a 2+2-week period followed by 2 weeks of suprasensory stimulation. Hereby rendering a stimulation test period of a total of 6 weeks (a permanent electrode is used).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18
* Patients who are psychologically stable and suitable for intervention and able to provide informed consent.
* Patients who are diagnosed with IBS-D or IBS-M according to the Rome III criteria
* Minimum average of 40 points in the symptom questionnaire evaluated at baseline

Exclusion Criteria:

* Overt bowel diseases including inflammatory bowel disease
* Pregnant or breast feeding
* Patients who are considered unable to follow the planned programme of the study, including mentally illness or physiological instability
* Patients who are on medication with known influence on gastrointestinal motility including those for thyroid disease, diabetes mellitus, celiac disease and neurological disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-09; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Cross sectional area | Change from baseline in cross sectional area at 6 weeks of stimulation
  Patients will be examined with Multimodal Stimulation using impedance planimetry measuring the cross sectional area before and after a standardised meal at baseline and at 6 weeks of stimulation

SECONDARY OUTCOMES:
Wall stiffness | Change from baseline in wall stiffness at 6 weeks of stimulation
  Patients will be examined with Multimodal Stimulation using impedance planimetry calculating the wall stiffness before and after a standardised meal at baseline and at 6 weeks of stimulation
Compliance | Change from baseline in compliance at 6 weeks of stimulation
  Patients will be examined with Multimodal Stimulation using impedance planimetry measuring the compliance before and after a standardised meal at baseline and at 6 weeks of stimulation
Cold | Change from baseline in cold tolerance at 6 weeks of stimulation
  Patients will be examined with Multimodal Stimulation using impedance planimetry measuring the cold tolerance before and after a standardised meal at baseline and at 6 weeks of stimulation
Heat | Change from baseline in heat tolerance at 6 weeks of stimulation
  Patients will be examined with Multimodal Stimulation using impedance planimetry measuring the heat tolerance before and after a standardised meal at baseline and at 6 weeks of stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Janne Fassov, PhD, Principal Investigator — Surgical Research Unit, Department of Surgery P, Aarhus University Hospital
Locations (1):
- Surgical Research Unit, Department of Surgery P, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided